CLINICAL TRIAL: NCT01773876
Title: Micafungin Versus Placebo in the Nosocomial Sepsis in Patients Multi-colonized With Candida, Randomized Controlled Trial
Brief Title: Empirical Antifungal Treatment in ICUS
Acronym: EMPIRICUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1126; 2011-005451-14 (Other: EudraCT number)
Record Dates: First submitted 2013-01-14; First posted 2013-01-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Invasive Candidiasis
Keywords: survival without proven invasive candidiasis; effectiveness; micafungin versus placebo; pharmacokinetic; pharmacodynamic; tolerance
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Micafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micafungin (Active Comparator): MYCAMINE 100 mg intravenous an injection of 24 hours
  Interventions: Drug: Micafungin
- PLACEBO (Placebo Comparator): 0.9% sodium chlorides 100ml infusion
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Micafungin — MYCAMINE 100 mg intravenous 100 mg of powder reconstituted in a 100 ml infusion bag of sodium chloride 0.9%
  infusion over 24 hours for 14 days discontinuation of treatment if proven invasive candidiasis
  Arms: Micafungin
Drug: PLACEBO — solution of sodium chloride 0.9% 100 ml for intravenous infusion infusion over 24 hours for 14 days discontinuation of placebo if proven invasive candidiasis
  Arms: PLACEBO

SUMMARY:
Invasive Candida infections are burdened with a high mortality rate and is very common in intensive care units. This study aims to evaluate the efficacy of empirical treatment with micafungin in adult patients with suspected invasive candidiasis.

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind parallel groups comparing adult patients with suspected invasive candidiasis input from a 14-day empirical treatment with micafungin (MYCAMINE 100 mg) with placebo on survival without invasive candidiasis in 28 days after initiation of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Persistent sepsis without documented invasive candidiasis:

systemic inflammatory response syndrome (SIRS) presence of two signs on the 4 [temperature <36 ° C or> 38 ° C, heart rate> 90/min, respiratory rate> 20/min or PaCO2 <32 mmHg, leukocytosis> 12,000 / mm3, <4.000/mm3 or presence of circulating immature forms (> 10% of cells)] mechanical ventilation (intubation or tracheostomy) for over 4 days (96 hours) central line use of broad-spectrum antibacterial for more than 4 calendar days (96 hours) in the previous week presence of at least one extra-digestive site colonized by Candida sp. (Urine, mouth, throat, upper and lower respiratory tract, skin folds, and suction drains after surgery ...), not lower digestive tract, are not taken into account the positive samples of rectal swabs and / or stool cultures, absence of proven bacterial infections untreated no evidence of invasive fungal infections (positive blood culture, positive culture of a surgical site, deep biopsy with fungal) infection or mold according to the criteria of the group "fungal infection of the EORTC" organ failure

* Hospitalization in intensive care for over 5 days (120 hours)
* Giving a free, informed and in writing. In the absence of the person of trust or a family member (if present)consent to emergency possible.
* Receiving a social security system,
* Negative pregnancy test for patients of childbearing age

Exclusion Criteria:

* Proven invasive fungal infection (positive blood culture, positive culture of a surgical site, deep biopsy with fungal infection), including aspergillosis requiring antifungal therapy at the time of randomization
* Prognosis of less than 48 hours (for which the patient outcome will be fatal whatever treatment),
* Echinocandin antifungal treatment by more than one day or another antifungal for over 72 hours in the week before the inclusion visit,
* Allergy, hypersensitivity or known intolerance to echinocandins antifungal or any of the excipients of the drug
* Neutropenia (ANC <500/mm3)
* History of organ and bone marrow,
* Recent chemotherapy (less than 6 months)
* Systemic immunosuppressive therapy in progress, other than with corticosteroids at doses below 2 mg / kg / day of prednisolone or equivalent
* Participation in another interventional study in the same ICU stay or making treatment being evaluated within 28 days prior to randomization
* Any clinical investigator deems incompatible with the conduct of the study in acceptable security conditions
* Pregnant and lactating women,
* Adults subject to a legal protection measure
* Persons deprived of their liberty by a judicial or administrative decision, those hospitalized without consent, persons admitted to a health facility or social purposes other than research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2012-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
survival to 28 days without proven fungal infection (a fungal infection occurring within 48 hours after inclusion will be considered available for inclusion) | 28 days follow-up
  breakthrough infection defined as a proven infection occurs at least 48 hours after initiation of treatment Proven infection is considered purchased after enrollment if the first significant positive levy occurs after the 48 th hour after enrollment.

SECONDARY OUTCOMES:
pharmacokinetic parameters: estimated gross exposure indices: AUC, Cmax, Cmin | during 24 hours (between the two first infusions)
  Reports AUC / MIC and Cmax / MIC will be calculated
evaluation of tolerance | 3 months
  For all patients who received at least one dose of treatment:
  * number of adverse events reported after randomization up to 28 days, only death will count up to 3 months post-randomization (information on the long-term survival collected by telephone),
  * changes in the clinical examination, vital signs and laboratory results,
  * overall survival defined as the time from randomization to date of death from any cause.
  * Changes in liver function tests (bilirubin, ALT, AST, rate prothrombin, alkaline phosphatase) at the end of treatment and at the end study
pharmacodynamic parameters: potential serum biomarkers of treatment efficacy (PCR Candida,1,3 β-D-glucan,mannan antigenemia,anti-mannan,Procalcitonin (proCT)) | during 28 days
pharmacodynamic parameters: Early prognostic factors of response: J7 survival without proven invasive candidiasis | during 14 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis possible on all-cause mortality at day 28 (end of study) and J90 (3 months post-randomization) | during 90 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis can free survival antifungal treatment at day 28 | during 28 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis possible evolution of organ failure during the study | during 90 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis possible the use of mechanical ventilation during the study | during 90 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis possible evolution of the colonization index during study | during 90 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis possible changes in serum biomarkers (1-3 β-D-glucan, mannan antigenemia, anti-mannan Candida PCR) during the study | during 90 days
Evaluate the impact of empiric treatment with micafungin in patients with invasive candidiasis possible on the incidence of pneumonia acquired bacterial mechanical ventilation (VAP). | during 90 days

CONTACTS AND LOCATIONS:
Overall Officials: TIMSIT JFT Jean François, PU-PH, Principal Investigator — University Hospital, Grenoble
Locations (22):
- France (22):
  - Hospital Aix en Provence, Aix-en-Provence
  - Hospital University of Besançon, Besançon
  - University Hospital of Avicennes, Bobigny
  - Hospital University of Bordeaux, Bordeaux
  - Hospital University of Clermont Ferrand, Clermont-Ferrand
  - University Hospital of Beaujon, Clichy
  - University Hospital of Dijon, Dijon
  - Hospital of Draguignan, Draguignan
  - Hospital University of Grenoble, Grenoble
  - Departemental Hospital of Roche sur Yon, La Roche-sur-Yon
  - Hospital of Versailles, Le Chesnay
  - University Hospital Edouard Herriot, Lyon
  - Hospital University of Montpellier, Montpellier
  - Interegional Hospital André Grégoire, Montreuil
  - University Hospital Saint Louis, Paris
  - University Hospital of La Pitié Salpetrière, Paris
  - Hospital St Joseph, Paris
  - Hospital University of Bichat, Paris
  - Hospital of Pontoise, Pontoise
  - Hospital University of Reims, Reims
  - University Hospital of Saint Etienne, Saint-Etienne
  - University Hospital of Strasbourg, Strasbourg

REFERENCES:
- [Derived] Timsit JF, Azoulay E, Schwebel C, Charles PE, Cornet M, Souweine B, Klouche K, Jaber S, Trouillet JL, Bruneel F, Argaud L, Cousson J, Meziani F, Gruson D, Paris A, Darmon M, Garrouste-Orgeas M, Navellou JC, Foucrier A, Allaouchiche B, Das V, Gangneux JP, Ruckly S, Maubon D, Jullien V, Wolff M; EMPIRICUS Trial Group. Empirical Micafungin Treatment and Survival Without Invasive Fungal Infection in Adults With ICU-Acquired Sepsis, Candida Colonization, and Multiple Organ Failure: The EMPIRICUS Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1555-1564. doi: 10.1001/jama.2016.14655. PMID 27706483
- [Derived] Timsit JF, Azoulay E, Cornet M, Gangneux JP, Jullien V, Vesin A, Schir E, Wolff M. EMPIRICUS micafungin versus placebo during nosocomial sepsis in Candida multi-colonized ICU patients with multiple organ failures: study protocol for a randomized controlled trial. Trials. 2013 Nov 21;14:399. doi: 10.1186/1745-6215-14-399. PMID 24261608